CLINICAL TRIAL: NCT01587261
Title: Prospective Placebo-Controlled Double-Blinded Trial for High-Dose Vitamin C Administration During the Acute Resuscitative Phase of Severe Thermal Injuries
Brief Title: Vitamin C for Severe Thermal Injuries
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This potential study was held up at the level of the FDA as they wouldn't approve and IND for the dose of vitamin C we wanted to use.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRA2012
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Severe Thermal Injury, Greater Than 20% TBSA
Keywords: Burns; Vitamin C; Thermal Injury; Fluid Resuscitation
MeSH Terms: conditions — Burns | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Victims of severe thermal injury receiving placebo Lactated Ringers solution for the first 24 hours
  Interventions: Drug: Placebo
- Vitamin C (Experimental): Victims of severe thermal injury receiving high-dose vitamin C 66 mg/kg/hr for the first 24 hours
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — Treatment Group will receive a dose of 66 mg/kg/hr of ascorbic acid injection for 24 hours after injury
  Other Names: High Dose Ascorbic Acid
  Arms: Vitamin C
Drug: Placebo — Lactated Ringers solution will be given at a similar volume to what the treatment group will receive
  Other Names: LR
  Arms: Placebo

SUMMARY:
Animal and human data have supported the notion that administration of large doses of Vitamin C has beneficial effects on those subjects suffering from large burns. This effect may be due, in part, to the antioxidant and free-radical-scavenging properties of Vitamin C. These studies have demonstrated an improvement in urine output during resuscitation and reduced need for fluid volumes during resuscitation. In turn, these subjects demonstrated a reduction of wound edema, improved respiratory status (demonstrated by improvements in P:F ratios and reduced ventilator days), and no differences in terms of the possible complications of high-dose vitamin C administration between standard and treatment groups. The purpose of this study is to prospectively determine if Vitamin C can be safely used as an adjunctive treatment for patients suffering severe thermal injuries. High-dose vitamin C administered at a dose of 66mg/kg/hr during the acute phase of severe burn injuries will reduce fluid requirements in the first 48 hours after injury.

DETAILED DESCRIPTION:
Subjects presenting within 6 hours of a severe thermal injury, defined as greater than 20% of their total body surface area, or their family members will be approached on admission to Parkland Memorial Hospital and informed of the study. Those electing to participate in the study will be randomized to receive either high-dose vitamin C (66mg/kg/hr for the first 24 hours, this dosage is based on prior human studies) in addition to the standard resuscitation algorithm (as per the Parkland Formula) or to a control group receiving only the standard resuscitation algorithm. These subjects will then be followed during their hospital course for fluid requirements, urine output, infectious complication rates, liver/renal failure rates, abdominal compartment syndrome rates, and outcomes such as ICU days, total hospital days, and mortality. All adverse events will be monitored by a data safety monitoring board. Currently this is a planned pilot study with a future multi-center study planned based on the results of the pilot. These studies will help determine if high-dose vitamin C can be a safe adjunct to acute fluid resuscitation in severely burned patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects presenting with second and/or third degree burns exceeding 20% total body surface area but not greater than 75% TBSA
2. Age between 18 and 65 years of age
3. Subject has provided full written informed consent prior to the performance of any study-related treatment or procedure

Exclusion Criteria:

1. Subjects presenting more than 6 hours from the estimated time of injury
2. Known inclusion in another interventional clinical trial
3. Subjects with known significant comorbidities (Congestive Heart Failure, Myocardial Infarction within 6 months of admission, Chronic Obstructive Pulmonary Disease, Chronic Kidney Disease or Renal Impairment)
4. Pregnant Subjects
5. Prisoners or Subjects Under Arrest
6. Subjects younger than 18 years of age or older than 65 years of age
7. Subjects with Baux Scores (Age plus % TBSA) greater than 120 (describing a non-survivable injury)
8. Subjects with any known allergy to components included in injectable ascorbic acid
9. Subjects with significant trauma burden (ISS > 15), including any open fracture, intracranial hemorrhage, or significant intra-abdominal injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Fluid Volume Requirements during the resuscitative phase after severe burn | 24 hours
  Primary Outcome is to reduce fluid outcome requirements within the first 24 hours after severe thermal injury

SECONDARY OUTCOMES:
Days of Ventilator Support Required | Hospital Course, estimated 6 weeks
  Comparisons between cohorts as to the number of days of ventilator support will be measured
Incidence of Abdominal Compartment Syndrome | Hospital Course, estimated 6 weeks
Complication and infection rates in the Vitamin C group | Hospital Course, estimated 6 weeks
Incidence of Renal Failure | Hospital Course, estimated 6 weeks
  Incidence of renal failure between cohorts will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Kareem R AbdelFattah, MD, Principal Investigator — UT-Southwestern; Victoria Warren, RN, Study Director — UT-Southwestern
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States